CLINICAL TRIAL: NCT06348628
Title: Motivational Interviewing for Weight Loss in the Management of Non Alcoholic Fatty Liver Disease - A Randomized Controlled Trial
Brief Title: Motivational Interviewing in the Management of Non Alcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Madunil Anuk Niriella (Other)
Responsible Party: Sponsor-Investigator, Madunil Anuk Niriella, Professor in Gastroenterology, University of Kelaniya
Organization: University of Kelaniya (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P/38/04/2021
Record Dates: First submitted 2024-03-25; First posted 2024-04-05 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2024-04

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Motivational Interview; Randomized Controlled Trial
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Motivational Interview with Placebo (Experimental): Each participant receives a motivational interview session at the recruitment, 1, 3, 6 months.
  Simultaneously, They receive dietary, exercise and lifestyle advices.
  Interventions: Behavioral: Motivational Interview; Behavioral: Placebo
- Placebo (Placebo Comparator): Participants receive dietary, exercise and lifestyle advices at the recruitment, 1, 3 and 6 months
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Motivational Interview — 4 Motivational interviews within first 6 months
  Arms: Motivational Interview with Placebo
Behavioral: Placebo — Advices on standard of care treatment of NAFLD within first 6 months

SUMMARY:
The goal of this study is to assess if motivational counselling works to reduce the weight in participants with Non Alcoholic Fatty Liver Disease (NAFLD).

DETAILED DESCRIPTION:
Participants with NAFLD who meet inclusion and exclusion criteria and who give informed written consent, will be randomly assigned to the intervention and control group. Randomization will be done by using a random sequence generator with concealed allocation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years to 60 years
* Body Mass Index (BMI) is 25 kg/m^2 or more
* Newly diagnosed with NAFLD based on clinical history, ultrasound scan and laboratory values

Exclusion Criteria:

* Any medical condition that will significantly alter the weight eg: hypothyroidism, hyperthyroidism, Cushing disease
* Having moderate/severe depressive disorders or psychotic symptoms and or substance use disorders that would reduce their capacity to give consent and engage in Motivational interview
* Who are on drugs which will affect weight or mood/affect (eg: corticosteroids)
* Pregnancy or expecting to be conceive within the study period
* Having any health conditions that would impede engagement in physical activities
* Having any health conditions that would compromise the ability to follow the recommended dietary behaviors
* Concurrent involvement in another weight loss programme

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 231 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
Change in weight after 1 year compared to baseline | Baseline, 3 months, 6 months, 12 months
  Weight is measured using a digital scale
Change in Aspartate aminotransferase (AST) level and Alanine aminotransferase (ALT) level after 1 year compared to baseline | Baseline and 12 months
  Lower AST and ALT levels have a better outcome
Change in platelet count after 1 year compared to baseline | Baseline and 12 months
  Lower platelet count has a poor outcome
Change in waist circumference and hip circumference after 1 year compared to baseline | Baseline and 12 months
  The waist circumference is measured at the narrowest part of the waist. The hip circumference is measured at the widest part of the hips. Both are measured by using a measuring tape.
Change in total fat percentage and visceral fat percentage after 1 year compared to baseline | Baseline and 12 months
  Both are measured by impedance method.

SECONDARY OUTCOMES:
Change in motivation for weight loss after 1 year compared to baseline | Baseline, 12 months
  It is assessed using the validated self-report University of Rhode Island Change Assessment (URICA) scale. The minimum value is -2 and the maximum value is +14. a higher score means a better outcome while a lower score means a poor outcome.
Change in depression, anxiety and stress after 1 year compared to baseline | Baseline, 12 months
  It is assessed using the Depression, Anxiety and Stress Scale-21 (DASS-21). The minimum value for depression is 0 while maximum value is 28. A score more than 21 means severe depression. A minimum value for anxiety is 0 while maximum value is 20. A score more than 15 means severe anxiety. A minimum value for stress is 0 while maximum value is 34. A score more than 26 means severe stress.
Change in quality of life after 1 year compared to baseline | Baseline, 12 months
  It is assessed using the World Health Organization Quality of Life Brief (WHOQOL-BREF) version. The minimum value is 0 and the maximum value is 100. A lower score indicates poor quality of life while a higher score indicates a good quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Aruni Hapangama, MBBS, MDPsych, FRANZCP, Study Director — The Alfred Hospital, Melbourne, Victoria, Australia
Locations (1):
- Faculty of Medicine, University of Kelaniya, Ragama, Western Province, Sri Lanka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Younossi ZM, Stepanova M, Afendy M, Fang Y, Younossi Y, Mir H, Srishord M. Changes in the prevalence of the most common causes of chronic liver diseases in the United States from 1988 to 2008. Clin Gastroenterol Hepatol. 2011 Jun;9(6):524-530.e1; quiz e60. doi: 10.1016/j.cgh.2011.03.020. Epub 2011 Mar 25. PMID 21440669
- [Background] Niriella MA, Pathmeswaran A, De Silva ST, Kasturiratna A, Perera R, Subasinghe CE, Kodisinghe K, Piyaratna C, Rishikesawan V, Dassanayaka AS, De Silva AP, Wickramasinghe R, Takeuchi F, Kato N, de Silva HJ. Incidence and risk factors for non-alcoholic fatty liver disease: A 7-year follow-up study among urban, adult Sri Lankans. Liver Int. 2017 Nov;37(11):1715-1722. doi: 10.1111/liv.13478. Epub 2017 Jun 10. PMID 28544258
- [Background] Hu XY, Li Y, Li LQ, Zheng Y, Lv JH, Huang SC, Zhang W, Liu L, Zhao L, Liu Z, Zhao XJ. Risk factors and biomarkers of non-alcoholic fatty liver disease: an observational cross-sectional population survey. BMJ Open. 2018 Apr 5;8(4):e019974. doi: 10.1136/bmjopen-2017-019974. PMID 29626047
- [Background] Hagstrom H, Nasr P, Ekstedt M, Hammar U, Stal P, Hultcrantz R, Kechagias S. Fibrosis stage but not NASH predicts mortality and time to development of severe liver disease in biopsy-proven NAFLD. J Hepatol. 2017 Dec;67(6):1265-1273. doi: 10.1016/j.jhep.2017.07.027. Epub 2017 Aug 10. PMID 28803953
- [Background] Kawamura Y, Arase Y, Ikeda K, Seko Y, Imai N, Hosaka T, Kobayashi M, Saitoh S, Sezaki H, Akuta N, Suzuki F, Suzuki Y, Ohmoto Y, Amakawa K, Tsuji H, Kumada H. Large-scale long-term follow-up study of Japanese patients with non-alcoholic Fatty liver disease for the onset of hepatocellular carcinoma. Am J Gastroenterol. 2012 Feb;107(2):253-61. doi: 10.1038/ajg.2011.327. Epub 2011 Oct 18. PMID 22008893
- [Background] Sarwar R, Pierce N, Koppe S. Obesity and nonalcoholic fatty liver disease: current perspectives. Diabetes Metab Syndr Obes. 2018 Sep 25;11:533-542. doi: 10.2147/DMSO.S146339. eCollection 2018. PMID 30288073
- [Background] Schubel R, Nonnenmacher T, Sookthai D, Gonzalez Maldonado S, Sowah SA, von Stackelberg O, Schlett CL, Grafetstatter M, Nabers D, Johnson T, Kirsten R, Ulrich CM, Kaaks R, Kauczor HU, Kuhn T, Nattenmuller J. Similar Weight Loss Induces Greater Improvements in Insulin Sensitivity and Liver Function among Individuals with NAFLD Compared to Individuals without NAFLD. Nutrients. 2019 Mar 4;11(3):544. doi: 10.3390/nu11030544. PMID 30836637
- [Background] Vilar-Gomez E, Martinez-Perez Y, Calzadilla-Bertot L, Torres-Gonzalez A, Gra-Oramas B, Gonzalez-Fabian L, Friedman SL, Diago M, Romero-Gomez M. Weight Loss Through Lifestyle Modification Significantly Reduces Features of Nonalcoholic Steatohepatitis. Gastroenterology. 2015 Aug;149(2):367-78.e5; quiz e14-5. doi: 10.1053/j.gastro.2015.04.005. Epub 2015 Apr 10. PMID 25865049
- [Background] Centis E, Moscatiello S, Bugianesi E, Bellentani S, Fracanzani AL, Calugi S, Petta S, Dalle Grave R, Marchesini G. Stage of change and motivation to healthier lifestyle in non-alcoholic fatty liver disease. J Hepatol. 2013 Apr;58(4):771-7. doi: 10.1016/j.jhep.2012.11.031. Epub 2012 Nov 29. PMID 23201248
- [Background] Stewart KE, Haller DL, Sargeant C, Levenson JL, Puri P, Sanyal AJ. Readiness for behaviour change in non-alcoholic fatty liver disease: implications for multidisciplinary care models. Liver Int. 2015 Mar;35(3):936-43. doi: 10.1111/liv.12483. Epub 2014 Mar 10. PMID 24521540
- [Background] Ceccarini M, Borrello M, Pietrabissa G, Manzoni GM, Castelnuovo G. Assessing motivation and readiness to change for weight management and control: an in-depth evaluation of three sets of instruments. Front Psychol. 2015 May 11;6:511. doi: 10.3389/fpsyg.2015.00511. eCollection 2015. PMID 26029126
- [Background] Rodriguez-Cristobal JJ, Alonso-Villaverde C, Panisello JM, Trave-Mercade P, Rodriguez-Cortes F, Marsal JR, Pena E. Effectiveness of a motivational intervention on overweight/obese patients in the primary healthcare: a cluster randomized trial. BMC Fam Pract. 2017 Jun 20;18(1):74. doi: 10.1186/s12875-017-0644-y. PMID 28633627
- [Background] Gelli C, Tarocchi M, Abenavoli L, Di Renzo L, Galli A, De Lorenzo A. Effect of a counseling-supported treatment with the Mediterranean diet and physical activity on the severity of the non-alcoholic fatty liver disease. World J Gastroenterol. 2017 May 7;23(17):3150-3162. doi: 10.3748/wjg.v23.i17.3150. PMID 28533672
- [Background] Mazzotti A, Caletti MT, Brodosi L, Di Domizio S, Forchielli ML, Petta S, Bugianesi E, Bianchi G, Marchesini G. An internet-based approach for lifestyle changes in patients with NAFLD: Two-year effects on weight loss and surrogate markers. J Hepatol. 2018 Nov;69(5):1155-1163. doi: 10.1016/j.jhep.2018.07.013. Epub 2018 Oct 2. PMID 30290973